CLINICAL TRIAL: NCT01691339
Title: Safety and Immunogenicity Among Adults of Fluzone®, Influenza Virus Vaccines 2012-2013 Formulation (Intradermal and Intramuscular Route)
Brief Title: Study of Fluzone® Influenza Virus Vaccines 2012-2013 Formulation Among Adults.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRC50; U 1111-1124-8310 (Other: WHO)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Fluzone® (Influenza Virus Vaccine) 2012-2013 Formulation; Fluzone® High-Dose (Influenza Virus Vaccine) 2012-2013 Formulation; Trivalent Inactivated Influenza Vaccine; Fluzone® Intradermal (Influenza Virus Vaccine) 2012-2013 Formulation
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluzone vaccine (Group 1) (Experimental): Adults 18 to < 65 years of age randomized to receive one dose of Fluzone vaccine intramuscularly
  Interventions: Biological: Influenza Virus Vaccine: Fluzone® 2012-2013 Formulation
- Fluzone Intradermal vaccine (Group 2) (Experimental): Adults 18 to < 65 years of age randomized to receive one dose of Fluzone Intradermal vaccine intradermally
  Interventions: Biological: Influenza Virus Vaccine: Fluzone® Intradermal 2012-2013 Formulation
- Fluzone vaccine (Group 3) (Experimental): Adults ≥ 65 years of age randomized to receive one dose of Fluzone vaccine intramuscularly
  Interventions: Biological: Influenza Virus Vaccine: Fluzone® 2012-2013 Formulation
- Fluzone High-Dose Vaccine (Group 4) (Active Comparator): Adults ≥ 65 years of age randomized to receive one dose of Fluzone High-Dose vaccine intramuscularly
  Interventions: Biological: Influenza Virus Vaccine: Fluzone® High-Dose 2012-2013 Formulation

INTERVENTIONS:
Biological: Influenza Virus Vaccine: Fluzone® 2012-2013 Formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® (2012-2013 Formulation)
  Arms: Fluzone vaccine (Group 1)
Biological: Influenza Virus Vaccine: Fluzone® Intradermal 2012-2013 Formulation — 0.1 mL, Intradermal
  Other Names: Fluzone® Intradermal (2012-2013 Formulation)
  Arms: Fluzone Intradermal vaccine (Group 2)
Biological: Influenza Virus Vaccine: Fluzone® 2012-2013 Formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® (2012-2013 Formulation)
  Arms: Fluzone vaccine (Group 3)
Biological: Influenza Virus Vaccine: Fluzone® High-Dose 2012-2013 Formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® High-Dose (2012-2013 Formulation)
  Arms: Fluzone High-Dose Vaccine (Group 4)

SUMMARY:
The aim of this study is to evaluate the safety and immunogenicity of Fluzone vaccine (18 years to <65 years of age and ≥ 65 years of age), Fluzone Intradermal vaccine (18 years to <65 years of age), and Fluzone High-Dose vaccine (≥ 65 years of age).

Primary Objective:

* To describe the safety of the 2012 - 2013 formulation of Fluzone and Fluzone Intradermal vaccines in adults 18 to < 65 years of age and the safety of the 2012 - 2013 formulation of Fluzone and Fluzone High-Dose vaccines in adults ≥ 65 years of age.

Observational Objectives:

* To describe the immunogenicity of the 2012 - 2013 formulation of Fluzone and Fluzone Intradermal vaccines in adults 18 to < 65 years of age and the immunogenicity of the 2012 - 2013 formulation of Fluzone and Fluzone High-Dose vaccines in adults ≥ 65 years of age.
* To evaluate the compliance, in terms of immunogenicity, of each study vaccine (Fluzone, Fluzone Intradermal, and Fluzone High-Dose) in the applicable age group with the requirements of the Committee for Human Medicinal Products (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96.
* To submit remaining available sera from subjects given Fluzone vaccine to the Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support selection and recommendation of strains for subsequent years' influenza vaccines.

DETAILED DESCRIPTION:
Participants 18 to < 65 years of age will be randomized to receive a dose of either Fluzone or Fluzone Intradermal vaccine and participants ≥ 65 years of age will be randomized to receive a dose of Fluzone or Fluzone High-Dose vaccine. All participants will be followed up for safety and immunogenicity. The duration of participation in the trial will be approximately 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* History of serious adverse reaction to any influenza vaccine
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Prior vaccination with any 2012 - 2013 formulation of influenza vaccine
* Known systemic hypersensitivity to eggs, chicken proteins, latex, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone, Fluzone Intradermal, or Fluzone High-Dose vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information)
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine
* Personal history of Guillain-Barré syndrome
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, as reported by the subject
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol or drug addiction that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 100.4°F) on the day of vaccination. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- United States (4):
  - Boca Raton, Florida
  - South Miami, Florida
  - Council Bluffs, Iowa
  - Metairie, Louisiana

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 19 through 27 September 2012 at 4 clinic centers in the United States.
Pre-assignment Details: A total of 200 participants who met all of the inclusion and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- Fluzone® Vaccine (Group 1): Adults 18 to < 65 years of age received one dose of Fluzone vaccine intramuscularly
- Fluzone® Intradermal Vaccine (Group 2): Adults 18 to < 65 years of age received one dose of Fluzone Intradermal vaccine intradermally
- Fluzone® Vaccine (Group 3): Adults ≥ 65 years of age received one dose of Fluzone vaccine intramuscularly
- Fluzone® High-Dose Vaccine (Group 4): Adults ≥ 65 years of age received one dose of Fluzone High-Dose vaccine intramuscularly
Period: Overall Study
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4)
Started | 50 | 50 | 51 | 49
Completed | 50 | 50 | 51 | 49
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4) | Total
Number analyzed (Participants) | 50 | 50 | 51 | 49 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 0 | 0 | 100
  >=65 years | 0 | 0 | 51 | 49 | 100
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (13.6) | 40.5 (14.2) | 73.3 (5.7) | 72.2 (5.2) | 57.4 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 32 | 35 | 127
  Male | 19 | 21 | 19 | 14 | 73
Region of Enrollment [Number; unit: Participants]
  United States | 50 | 50 | 51 | 49 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With Fluzone® or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Solicited injection site: Pain, Erythema, Swelling, Induration, and Ecchymosis; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering.
  Grade 3 injection site: Pain - Significant, prevents daily activity; Erythema, Swelling, Induration, and Ecchymosis - >100 mm. Grade 3 systemic reactions: Fever ≥39.0°C; Headache, Malaise, Myalgia, and Shivering - significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4)
Number analyzed (Participants) | 50 | 50 | 51 | 49
Participants
  Injection site Pain | 12 | 20 | 12 | 19
  Grade 3 Injection site Pain | 0 | 0 | 0 | 0
  Injection site Erythema | 1 | 16 | 0 | 1
  Grade 3 Injection site Erythema | 0 | 0 | 0 | 0
  Injection site Swelling | 1 | 9 | 0 | 1
  Grade 3 Injection site Swelling | 0 | 0 | 0 | 0
  Injection site Induration | 1 | 4 | 0 | 1
  Grade 3Injection site Induration | 0 | 0 | 0 | 0
  Injection site Ecchymosis | 0 | 1 | 0 | 0
  Grade 3 Injection site Ecchymosis | 0 | 0 | 0 | 0
  Fever | 2 | 0 | 0 | 0
  Grade 3 Fever | 0 | 0 | 0 | 0
  Headache | 10 | 12 | 11 | 7
  Grade 3 Headache | 1 | 1 | 0 | 0
  Malaise | 11 | 11 | 10 | 7
  Grade 3 Malaise | 0 | 0 | 0 | 0
  Myalgia | 10 | 10 | 13 | 7
  Grade 3 Myalgia | 0 | 0 | 2 | 0
  Shivering | 4 | 4 | 4 | 3
  Grade 3 Shivering | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Geometric Mean Titers Against the Influenza Virus Antigens Following Vaccination With Fluzone® or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) up to Day 21 post-vaccination
Population: Geometric mean titers against the influenza virus antigens were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4)
Number analyzed (Participants) | 46 | 47 | 49 | 46
Titers
  A/H1N1 (Pre-vaccination; N = 46, 46, 49, 46) | 28.3 [17.5 to 45.6] | 30.7 [18.3 to 51.7] | 58.6 [37.5 to 91.6] | 81.8 [50.2 to 133]
  A/H1N1 (Post-vaccination; N = 46, 47, 49, 46) | 1068 [755 to 1512] | 1473 [955 to 2269] | 246 [177 to 343] | 369 [266 to 513]
  A/H3N2 (Pre-vaccination; N = 46, 46, 49, 46) | 29.1 [18.0 to 47.3] | 23.6 [14.3 to 39.0] | 68.5 [42.6 to 110] | 78.2 [50.2 to 122]
  A/H3N2 (Post-vaccination; N = 45, 47, 49, 46) | 460 [306 to 691] | 599 [369 to 971] | 264 [176 to 397] | 392 [266 to 578]
  B (Pre-vaccination; N = 46, 46, 49, 46) | 17.9 [13.0 to 24.6] | 20.9 [15.5 to 28.3] | 13.7 [10.5 to 17.7] | 18.7 [14.4 to 24.3]
  B (Post-vaccination; N = 45, 47, 49, 46) | 169 [131 to 218] | 129 [91.1 to 183] | 35.2 [25.8 to 48.1] | 60.1 [43.8 to 82.4]

3. Other Pre Specified Outcome: Number of Participants With Seroprotection Against Influenza Vaccine Antigens Before and Following Vaccination With Fluzone® or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay. Seroprotection was defined as a pre-vaccination or a post-vaccination titer ≥ 40 (l/dil).
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Seroprotection against influenza vaccine antigens were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4)
Number analyzed (Participants) | 46 | 47 | 49 | 46
Participants
  A/H1N1 (Pre-vaccination; N = 46, 46, 49, 46) | 22 [32.9 to 63.1] | 23 [34.9 to 65.1] | 32 [50.4 to 78.3] | 33 [56.5 to 84.0]
  A/H1N1 (Post-vaccination; N = 46, 47, 49, 46) | 46 [92.3 to 100.0] | 46 [88.7 to 99.9] | 49 [92.7 to 100.0] | 45 [88.5 to 99.9]
  A/H3N2 (Pre-vaccination; N = 46, 46, 49, 46) | 22 [32.9 to 63.1] | 15 [19.5 to 48.0] | 33 [52.5 to 80.1] | 31 [52.0 to 80.5]
  A/H3N2 (Post-vaccination; N = 45, 47, 49, 46) | 44 [88.2 to 99.9] | 45 [85.5 to 99.5] | 46 [83.1 to 98.7] | 45 [88.5 to 99.9]
  B (Pre-vaccination; N = 46, 46, 49, 46) | 9 [9.4 to 33.9] | 15 [19.5 to 48.0] | 8 [7.3 to 29.7] | 13 [16.0 to 43.5]
  B (Post-vaccination; N = 45, 47, 49, 46) | 45 [92.1 to 100.0] | 40 [71.7 to 93.8] | 26 [38.3 to 67.5] | 33 [56.5 to 84.0]

4. Other Pre Specified Outcome: Number of Adult Participants With Seroconversion to Influenza Virus Vaccine Antigens Following Vaccination With Fluzone® or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay. Seroconversion was defined as either a pre-vaccination titer < 10 (1/dil) and a post-vaccination titer ≥ 40 (1/dil), or a pre-vaccination titer ≥ 10 (1/dil) and a ≥ 4-fold increase in post-vaccination titer.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Seroconversion to the influenza virus vaccine antigens was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4)
Number analyzed (Participants) | 46 | 47 | 49 | 46
Participants
  A/H1N1 (N = 46, 46, 49, 46) | 43 [82.1 to 98.6] | 43 [82.1 to 98.6] | 21 [28.8 to 57.8] | 26 [41.1 to 71.1]
  A/H3N2 (N = 45, 46, 49, 46) | 34 [60.5 to 87.1] | 39 [71.1 to 93.7] | 19 [25.2 to 53.8] | 28 [45.4 to 74.9]
  B (N = 45, 46, 49, 46) | 36 [65.4 to 90.4] | 33 [56.5 to 84.0] | 13 [14.9 to 41.1] | 16 [21.4 to 50.2]

5. Other Pre Specified Outcome: Number of Participants With Influenza Antibody Titers of <1:10 Before and Following Vaccination With Fluzone® or Fluzone® Intradermal or Fluzone® High-Dose Vaccine
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay to determine pre-vaccination and post-vaccination titers of <1:10.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Antibody responses to the influenza vaccine antigens were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® Vaccine (Group 1) | Fluzone® Intradermal Vaccine (Group 2) | Fluzone® Vaccine (Group 3) | Fluzone® High-Dose Vaccine (Group 4)
Number analyzed (Participants) | 46 | 47 | 49 | 46
Participants
  A/H1N1 (Pre-vaccination; N = 46, 46, 49, 46) | 18 [25.1 to 54.6] | 17 [23.2 to 52.5] | 6 [4.6 to 24.8] | 6 [4.9 to 26.3]
  A/H1N1 (Post-vaccination; N = 46, 47, 49, 46) | 0 [0 to 7.7] | 1 [0.1 to 11.3] | 0 [0 to 7.3] | 0 [0 to 7.7]
  A/H3N2 (pre-vaccination; N = 46, 46, 49, 46) | 17 [23.2 to 52.5] | 19 [27.0 to 56.8] | 6 [4.6 to 24.8] | 2 [0.5 to 14.8]
  A/H3N2 (Post-vaccination; N = 45, 47, 49, 46) | 0 [0 to 7.9] | 1 [0.1 to 11.3] | 0 [0 to 7.3] | 0 [0 to 7.7]
  B (Pre-vaccination; N = 46, 46, 49, 46) | 12 [14.3 to 41.1] | 9 [9.4 to 33.9] | 17 [21.7 to 49.6] | 13 [16.0 to 43.5]
  B (Post-vaccination; N = 45, 47, 49, 46) | 0 [0 to 7.9] | 1 [0.1 to 11.3] | 4 [2.3 to 19.6] | 1 [0.1 to 11.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Groups:
- Fluzone Vaccine (Group 1): 'Adults 18 to < 65 years of age received one dose of Fluzone vaccine intramuscularly'
- Fluzone Intradermal Vaccine (Group 2): Adults 18 to < 65 years of age received one dose of Fluzone Intradermal vaccine intradermally
- Fluzone Vaccine (Group 3): Adults ≥ 65 years of age received one dose of Fluzone vaccine intramuscularly
- Fluzone High-Dose Vaccine (Group 4): Adults ≥ 65 years of age received one dose of Fluzone High-Dose vaccine intramuscularly
Arm/Group | Fluzone Vaccine (Group 1) | Fluzone Intradermal Vaccine (Group 2) | Fluzone Vaccine (Group 3) | Fluzone High-Dose Vaccine (Group 4)
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 2/51 | 0/49
Other Adverse Events (participants affected / at risk) | 12/50 | 20/50 | 13/51 | 19/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Vaccine (Group 1) (N=50) | Fluzone Intradermal Vaccine (Group 2) (N=50) | Fluzone Vaccine (Group 3) (N=51) | Fluzone High-Dose Vaccine (Group 4) (N=49)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Vaccine (Group 1) (N=50) | Fluzone Intradermal Vaccine (Group 2) (N=50) | Fluzone Vaccine (Group 3) (N=51) | Fluzone High-Dose Vaccine (Group 4) (N=49)
Injection site Pain (General disorders) | 12 (12) | 20 (20) | 12 (12) | 19 (19)
Injection site Erythema (General disorders) | 1 (1) | 16 (16) | 0 (0) | 1 (1)
Injection site Swelling (General disorders) | 1 (1) | 9 (9) | 0 (0) | 1 (1)
Injection site Induration (General disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Headache (General disorders) | 10 (10) | 12 (12) | 11 (11) | 7 (7)
Malaise (General disorders) | 11 (11) | 11 (11) | 10 (10) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (10) | 13 (13) | 7 (7)
Shivering (General disorders) | 4 (4) | 4 (4) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications